CLINICAL TRIAL: NCT06891053
Title: Studio TIARA: Alessitimia ed Emicrania Cronica
Acronym: TIARA
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Sanitaria Locale di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: Asl22.Neuro.22.01
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Migraine; Alexithymia
MeSH Terms: conditions — Migraine Disorders; Affective Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosis of episodic migraine without or with aura, chronic migraine, and/or MOH: Female patients, aged 12-65 years, diagnosed with episodic migraine without or with aura, chronic migraine, and/or MOH according to the criteria of ICHD-3 2018

SUMMARY:
The aim of this observational, cross-sectional study is to investigate the relationship between alexithymia and migraine frequency (considering alexithymia a condition that can influence the severity of the clinical phenotype of migraine, favoring its chronicization), in an analysis adjusted for psychiatric comorbidity (for anxiety and depression, potentially influencing migraine chronicization) and for personalogical factor represented by apathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of episodic migraine with or without aura, chronic migraine and/or MOH according to ICHD-3 2018 criteria;
* Patients aged 12-65 years;
* Female patients

Exclusion Criteria:

* Ongoing major depressive episode;
* Comorbidities for major internal diseases (hepatopathy, nephropathy, heart failure, etc.);
* Alcohol or substance abuse disorder (eoin, cocaine, cannabis, hallucinogens);
* Language barrier;
* Low cultural/cognitive level;
* No informed consent.

Ages: 12 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female patients, aged 12-65 years, diagnosed with episodic migraine with or without aura, chronic migraine and/or MOH according to ICHD-3 2018 criteria
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of alexithymia | In 3 periods of 30 days each (3 months), which make up the 90-day observation time interval
  Independent variable measured as a score on the TAS-20 scale
Migraine frequency | In 3 periods of 30 days each (3 months), which make up the 90-day observation time interval

SECONDARY OUTCOMES:
Number of "drug days" in patients diagnosed with MOH | In 3 periods of 30 days each (3 months), which make up the 90-day observation time interval
Degree of alessithymia in patients diagnosed with MOH | In 3 periods of 30 days each (3 months), which make up the 90-day observation time interval

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Rota, Principal Investigator — Azienda Sanitaria Locale di Alessandria (ASL AL)
Locations (1):
- Azienda Sanitaria Locale di Alessandria (ASL AL), Alessandria, Italy, Italy

IPD SHARING:
Plan to Share IPD: No